CLINICAL TRIAL: NCT03287349
Title: Genomic Assessment of Patients With Severe Radiation Reactions
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 16-004880
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-07

CONDITIONS: Radiation; Reaction
MeSH Terms: interventions — Blood Specimen Collection; Moire Topography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with severe reactions to radiation: Two 12.5 mL blood draws and photograph of severe reaction, and autoimmune testing in patients without prior testing.
  Interventions: Other: Blood draw; Other: Photograph; Diagnostic Test: Autoimmune testing

INTERVENTIONS:
Other: Blood draw — Two 12.5 mL blood draws
Other: Photograph — Photograph of severe reaction, will be anonymized
Diagnostic Test: Autoimmune testing — Autoimmune testing in patients without prior testing

SUMMARY:
Determine an underlying etiology behind unexpectedly severe reactions to radiation by blood draw.

ELIGIBILITY:
Inclusion Criteria:

* Weigh at least 110 pounds
* Healthy

Exclusion Criteria:

- Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adults with severe reactions to radiation treatment
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Whole exome sequencing | baseline
  Investigate genes potentially responsible for severe radiation reactions by getting blood draws.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Corbin, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials